CLINICAL TRIAL: NCT00579124
Title: CHP 834 Unrelated and Partially Matched Related Donor Peripheral Stem Cell Transportation With the CliniMACs Device for T and B Cell Depletion
Brief Title: CHP 834 Unrelated and Partially Matched Related Donor Peripheral Stem Cell Transportation for T and B Cell Depletion
Acronym: CliniMACs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Nancy Bunin, BMT Medical Director, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-004222
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2024-01-18 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Immunodeficiencies
Keywords: Blood and Marrow Transplant; T cell Depletion; Unrelated; Related; Donor
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. CliniMACS CD3+/CD19+ depletion (Other): * 6/6 or 8/8 matched (fully matched)
  * 1 antigen or allele mismatched (mismatch at A or B or DRB1)
  * 2 antigen or allele mismatched (mismatch ONLY at A and B but NOT at DRB1 plus either A or B).
  Patients will receive grafts that have undergone CD3+ and CD19+ depletion. The CD3(-) fraction will be infused.
  Interventions: Device: CliniMACs
- 2. CliniMACS CD3+/CD19+ depletion (Other): Stratum 2. CliniMACS CD3+/CD19+ depletion:
  * Haploidentical match
  * 2 antigen and/or allele mismatched where one of the mismatches includes DRB1
  For patients in Stratum 2 we will perform CD3+ (T cell) and CD19+ (B cell) depletion. There will be no T cell add back in this stratum.
  Interventions: Device: CliniMACs

INTERVENTIONS:
Device: CliniMACs — T and B Cell depletion
  Other Names: T and B Cell depletion; DONOR PERIPHERAL STEM CELL TRANSPLANTATION

SUMMARY:
This is a pilot study with 2 strata to evaluate engraftment and graft vs. host disease (GVHD) in patients receiving unrelated or partially matched related donor peripheral stem cells using the CliniMACS system to positively deplete T cells to prevent severe GVHD. Feasibility will be tested, focusing on engraftment, treatment-related mortality (with a specific focus on interstitial pneumonitis) and severe GVHD.

DETAILED DESCRIPTION:
PRIMARY HYPOTHESIS: T cell depletion utilizing the CliniMACS device will allow more precise, specific and controlled graft engineering of peripheral blood stem cells from unrelated and partially matched related donors without an increase in relapse or graft rejection and grade III or IV acute graft vs. host disease (GVHD).

SECONDARY HYPOTHESIS: Use of the CliniMACS device will allow defined levels of T cell depletion to reflect the risk of severe GVHD in the donor/recipient pair.

Thus, patients with a relatively lower risk of severe GVHD will be assigned to Stratum 1 and receive a graft with lesser T cell depletion and a defined level of reinfused T cells. Patients with higher risk of severe GVHD or for whom there is no perceived clinical benefit of GVHD will be assigned to Stratum 2 and receive a more T cell-depleted graft.

Conditioning of the patient (except immunodeficiencies) includes :

* Thiotepa 5 mg/kg days for 2 days
* Cyclophosphamide 60 mg/kg days for 2 days
* Total body irradiation 200 cGy given twice a day for 3 days

Following conditioning patient's will receive stem cells that have been processed using the CliniMACS device. This processing is done in the stem cell laboratory at The Children's Hospital of Philadelphia. The Stem Cell Lab is accredited by the Foundation for the Accreditation of Cellular Therapy (FACT) and maintain complete standard operating procedures (SOP's) and procedure records.

Processing of cells using the CliniMACS will occur in accordance with the Investigator Brochure and Technical Manual following the laboratory SOPs and using aseptic technique. The CHOP Stem Cell Lab has extensive prior experience with automated cell processing technologies, including the CellPro Ceprate device and the Isolex 300i.

ELIGIBILITY:
Inclusion Criteria:

As of October 2014 this study closed enrollment to malignant diseases. This study remains open to:

Non-malignant diseases:

1. Bone marrow failure, including severe aplastic anemia
2. Immunodeficiencies

Exclusion Criteria:

1. Patients who have had prior stem cell transplant (SCT) and bone marrow transplant (BMT) are excluded for study enrollment.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 93 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Bunin, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Seif AE, Li Y, Monos DS, Heidemann SC, Aplenc R, Barrett DM, Casper JT, Freedman JL, Grupp SA, Margolis DA, Olson TS, Teachey DT, Keever-Taylor CA, Wang Y, Talano JM, Bunin NJ. Partially CD3+-Depleted Unrelated and Haploidentical Donor Peripheral Stem Cell Transplantation Has Favorable Graft-versus-Host Disease and Survival Rates in Pediatric Hematologic Malignancy. Biol Blood Marrow Transplant. 2020 Mar;26(3):493-501. doi: 10.1016/j.bbmt.2019.11.022. Epub 2019 Nov 22. PMID 31765697
- See also: Partially CD3+ -Depleted Unrelated and Haploidentical Donor Peripheral Stem Cell Transplantation Has Favorable Graft-versus-Host Disease and Survival Rates in Pediatric Hematologic Malignancybiol — http://doi.org/10.1016/j.bbmt.2019.11.022

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. CliniMACS CD3+/CD19+ Depletion: * 6/6 or 8/8 matched (fully matched)
  * 1 antigen or allele mismatched (mismatch at A or B or DRB1)
  * 2 antigen or allele mismatched (mismatch ONLY at A and B but NOT at DRB1 plus either A or B).
  Patients will receive grafts that have undergone CD3+ and CD19+ depletion. The CD3(-) fraction will be infused.
  CliniMACs: T and B Cell depletion
- 2. CliniMACS CD3+/CD19+ Depletion: Stratum 2. CliniMACS CD3+/CD19+ depletion:
  * Haploidentical match
  * 2 antigen and/or allele mismatched where one of the mismatches includes DRB1
  For patients in Stratum 2 we will perform CD3+ (T cell) and CD19+ (B cell) depletion. There will be no T cell add back in this stratum.
  CliniMACs: T and B Cell depletion
Period: Overall Study
Arm/Group | 1. CliniMACS CD3+/CD19+ Depletion | 2. CliniMACS CD3+/CD19+ Depletion
Started | 87 | 6
Completed | 82 | 6
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stratum 1: Stratum 1. CliniMACS CD3+/CD19+ depletion: Patients with donors with the following levels of matching:
  * 6/6 or 8/8 matched (fully matched)
  * 1 antigen or allele mismatched (mismatch at A or B or DRB1)
  * 2 antigen or allele mismatched (mismatch ONLY at A and B but NOT at DRB1 plus either A or B).
- Stratum 2: * Haploidentical match
  * 2 antigen and/or allele mismatched where one of the mismatches includes DRB1
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 87 | 6 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 80 | 6 | 86
  Between 18 and 65 years | 7 | 0 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 12 [1 to 21] | 0.5 [0 to 1] | 12 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 0 | 44
  Male | 43 | 6 | 49
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 6 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Engraftment
Description: Successful engraftment will be whether subjects have achieved an absolute neutrophil count (ANC) >500 and platelet count >20 x 109/l by 100 days after transplant
Time Frame: 100 days Post Transplant
Measure: Count of Participants; unit: Participants
Groups:
- Stratum 2: Patients with donors with the following levels of matching:
  * Haploidentical match
  * 2 antigen and/or allele mismatched where one of the mismatches includes DRB1
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 87 | 5
Participants | 87 | 5

ADVERSE EVENTS:
Groups:
- AEs for Total Number of Participants: Stratum 1: this group is total subject count evaluated for AE results in Stratum 1
- AEs for Total Number of Participants: Stratum 2: this group is total subject count evaluated for AE results in Stratum 2
Arm/Group | AEs for Total Number of Participants: Stratum 1 | AEs for Total Number of Participants: Stratum 2
All-Cause Mortality (participants affected / at risk) | 0/87 | 2/6
Serious Adverse Events (participants affected / at risk) | 6/87 | 2/6
Other Adverse Events (participants affected / at risk) | 0/87 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEs for Total Number of Participants: Stratum 1 (N=87) | AEs for Total Number of Participants: Stratum 2 (N=6)
Non-relapsed mortality (General disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No